CLINICAL TRIAL: NCT05851976
Title: Duloxetine for Patients With Low Back Pain Who Fail to Improve With Oral NSAIDs. A Randomized Placebo-controlled Exploratory Study
Brief Title: Duloxetine for LBP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-14971
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Back Pain, Low
MeSH Terms: conditions — Low Back Pain | interventions — Naproxen; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naproxen + duloxetine (Experimental)
  Interventions: Drug: Naproxen; Drug: Duloxetine
- Naproxen + placebo (Placebo Comparator)
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Naproxen — Naproxen 500mg twice daily for 16 days
Drug: Duloxetine — Duloxetine 60mg daily for 14 days
  Arms: Naproxen + duloxetine

SUMMARY:
This research study will help determine whether a medication called duloxetine can improve back pain. It is well documented that many participants who come to the ER with acute low back pain still have low back pain 3 months later. The investigator team will attempt to determine whether duloxetine can help prevent this.

DETAILED DESCRIPTION:
Participants will be eligible to take duloxetine/placebo if insufficient relief of pain after using naproxen for 48 hours has been reported.

ELIGIBILITY:
Inclusion Criteria:

* Present to Emergency Department (ED) primary for management of LBP, defined as pain originating between the lower border of the scapulae and the upper gluteal folds. Flank pain, that is pain originating from tissues lateral to the paraspinal muscles, will not be included.
* Musculoskeletal etiology of low back. Patients with non-musculoskeletal etiologies such as urinary tract infection, ovarian cysts, or influenza like illness will be excluded. The primary clinical diagnosis, at the conclusion of the ED visit, must be a diagnosis consistent with non-traumatic, non-radicular, musculoskeletal LBP.
* Patient is to be discharged home. Patients admitted to the hospital are more likely to be treated with parenteral medication and therefore are not appropriate for this study.
* Age 18-64 Enrollment will be limited to adults younger than 65 years because of the increased risk of adverse medication effects in older patients.
* Non-radicular pain. Patients will be excluded if the pain radiates below the gluteal folds in a radicular pattern.
* Pain duration <2 weeks (336 hours).
* Prior to the acute attack of LBP, back pain cannot occur more frequently than once per week.
* Functionally impairing back pain: A baseline score of > 5 on the Roland-Morris Disability Questionnaire

Exclusion Criteria:

* Not available for follow-up
* Pregnant or breast-feeding
* Chronic pain syndrome defined as moderate or severe pain anywhere in their body on >= 50% of days for at least three months
* Allergic to or intolerant of investigational medications
* Contra-indications to non-steroidal anti-inflammatory drugs:

  1. history of hypersensitivity to NSAIDs or aspirin
  2. active or history of peptic ulcer disease, chronic dyspepsia, or active or history of gastrointestinal bleed
  3. Severe heart failure (NYHA 2 or worse)
  4. uncontrolled blood pressure (>160/100)
  5. Glomerular Filtration Rate (GFR) <60ml/min
  6. Current use of anti-coagulants
  7. cirrhosis or acute hepatitis
* Contra-indication to duloxetine:

  1. alcohol use disorder
  2. chronic liver disease
  3. chronic kidney disease
  4. glaucoma
  5. Active use of medication for depression
  6. Score > 10 on the Patient Health Questionnaire (PHQ-9) screening instrument or thoughts of suicide, symptoms of feeling down, depressed, or hopeless

PHQ9 score >4. Now we would like to exclude patients with a PHQ9 score >10 or symptoms of feeling down, depressed, or hopeless

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with moderate or severe Low Back Pain (LBP) | 16 days, 42 days and 84 days after ED discharge
  An ordinal pain scale ("severe", "moderate", "mild", or "none") will be used to assess LBP. Study participants will be asked to describe their worst back pain over the previous 24 hours. The number of patients reporting with "Moderate" or "Severe" pain will be summarized by study arm.

SECONDARY OUTCOMES:
Number of Participants experiencing LBP based on the Roland Morris Disability Questionnaire (RMDQ) | 9 days, 16 days, 23 days, and 42 days after Emergency Department (ED) discharge
  The Roland Morris Disability Questionnaire (RMDQ) will be used to assess the number of participants experiencing LBP over the prior 24-hour period. Items on the 24-item functional scale are scored 0 if left blank or 1 if endorsed, for a total Roland Morris score ranging from 0-24. Group scores will be summarized by study arm using basic descriptive statistics. Higher scores represent higher levels of pain-related disability.
Frequency of LBP | 9 days, 16 days, 23 days, and 42 days after ED discharge
  Frequency of LBP will be assessed by the response to the question, "Over the last 24 hours, how often were you in pain?" Response options on the questionnaire will be limited to "Not at all," "Rarely," " Sometimes," "Usually," or "Always." Since LBP symptomatology is quite variable, this question will help determine the burdensomeness of LBP on the patient's daily life. Responses will be summarized and reported by study arm.
Number of visits to a healthcare provider | 9 days, 16 days, 23 days, and 42 days after ED discharge
  The number of visits to any healthcare provider since the prior visit will be summarized by study arm using basic descriptive statistics by study arm. Visits can include any visit to a primary, secondary, or tertiary healthcare provider.
The number of patients experiencing Depressive Symptoms | 9 days, 16 days, 23 days, and 42 days after ED discharge
  Number of participants demonstrating depressive symptoms over the prior 2 week period will be assessed using the 9-item Patient Health Questionnaire (PHQ-9). The PHQ-9 is an instrument used for the screening, diagnosing, monitoring, and measuring the severity of depression. Responses to the 9 questions are based on 4-point Likert-like scale ranging from 0 ("Not at all") to 3 ("Nearly every day") for an overall possible scoring range of 0-27. Higher scores are associated with increased depressive symptoms. Scores will be summarized by study arm using basic descriptive statistics.
The number of patients reporting Satisfaction with treatment | 9 days, 16 days, 23 days, and 42 days after ED discharge
  The number of patients reporting satisfaction will be assessed by the response to the question, "The next time you go to the ER with LBP back do you want to get the same combination of medications?" Responses will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No